CLINICAL TRIAL: NCT01232335
Title: Symbicort Turbuhaler 30/60 Specific Clinical Experience Investigation for Long-term Use
Brief Title: Symbicort Turbuhaler 30/60 Specific Clinical Experience Investigation
Acronym: ENSURE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D589IC00001
Record Dates: First submitted 2010-10-31; First posted 2010-11-02 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Bronchial Asthma
Keywords: bronchial asthma; Symbicort; long term use,
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to confirm the safety profile for long term treatment and maximize doses and the control status on bronchial asthma in daily clinical usage

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Symbicort for the first time possibly at the higher dose due to bronchial asthma

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Symbicort for the first time due to bronchial asthma
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Range of one year

SECONDARY OUTCOMES:
The level of asthma control under long-term use | At the end of 24 weeks
The level of asthma control under long-term use | At the end of one year

CONTACTS AND LOCATIONS:
Overall Officials: Yoshida Shigeru, Study Director — AstraZeneca
Locations (47):
- Japan (47):
  - Research Site, Aichi, Japan
  - Research Site, Akita, Japan
  - Research Site, Aomori, Japan
  - Research Site, Chiba, Japan
  - Research Site, Ehime, Japan
  - Research Site, Fukui, Japan
  - Research Site, Fukuoka, Japan
  - Research Site, Fukushima, Japan
  - Research Site, Gifu, Japan
  - Research Site, Gunma, Japan
  - Research Site, Hiroshima, Japan
  - Research Site, Hokkaido, Japan
  - Research Site, Hyōgo, Japan
  - Research Site, Ibaraki, Japan
  - Research Site, Ishikawa, Japan
  - Research Site, Kagawa, Japan
  - Research Site, Kagoshima, Japan
  - Research Site, Kanagawa, Japan
  - Research Site, Kochi, Japan
  - Research Site, Kumamoto, Japan
  - Research Site, Kyoto, Japan
  - Research Site, Mie, Japan
  - Research Site, Miyagi, Japan
  - Research Site, Miyazaki, Japan
  - Research Site, Nagano, Japan
  - Research Site, Nagasaki, Japan
  - Research Site, Nara, Japan
  - Research Site, Niigata, Japan
  - Research Site, Numakunai, Japan
  - Research Site, Okayama, Japan
  - Research Site, Okinawa, Japan
  - Research Site, Osaka, Japan
  - Research Site, Ōita, Japan
  - Research Site, Saga, Japan
  - Research Site, Saitama, Japan
  - Research Site, Shiga, Japan
  - Research Site, Shimane, Japan
  - Research Site, Shizuoka, Japan
  - Research Site, Tochigi, Japan
  - Research Site, Tokushima, Japan
  - Research Site, Tokyo, Japan
  - Research Site, Tottori, Japan
  - Research Site, Toyama, Japan
  - Research Site, Wakayama, Japan
  - Research Site, Yamagata, Japan
  - Research Site, Yamaguchi, Japan
  - Research Site, Yamanashi, Japan